CLINICAL TRIAL: NCT04061408
Title: A Phase II Pilot Study of Fractionated Stereotactic Radiotherapy(FSRT) in Breast Cancer Patients With 1 to 10 Brain Metastases
Brief Title: FSRT in Breast Cancer Patients With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-BC009
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Brain Metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FSRT (Experimental): 3 to 5 fractions and 8Gy per fraction will be used for breast cancer patients with 1-10 brain metastases based on the lesion number and volume.
  Interventions: Radiation: Fractionated stereotactic radiotherapy(FSRT)

INTERVENTIONS:
Radiation: Fractionated stereotactic radiotherapy(FSRT) — 3 to 5 fractions and 8Gy per fraction will be used for breast cancer patients with 1-10 brain metastases based on the lesion number and volume.

SUMMARY:
Brain metastasis accounted for 10-15% of all breast cancer patients and even higher in patients with triple negative and HER2 overexpressed subtype. Stereotactic radiation is the standard option for patients with 1-4 brain metastases. Among patients with 1-4 brain metastases, many studies suggest that stereotactic radiation results in fewer neurologic side effects than whole brain radiation. Also, several studies had demonstrated that 5-10 lesions had similar overall survival by using whole brain radiotherapy or stereotactic radiotherapy. Fractionated stereotactic radiotherapy(FSRT) is increasingly administered in the brain metastatic patients and retrospective studies had shown that FSRT had better local control and lower brain radiation necrosis than single fraction stereotactic radiation. Therefore, In this study, we explore to treat 1-10 brain metastasis lesion in breast cancer patients with FSRT.

DETAILED DESCRIPTION:
Breast cancer patients with 1-10 brain metastasis will be treated with FSRT for brain metastasis. 3 to 5 fractions and 8Gy per fraction will be used for these patients based on the lesion number and volume.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HER2 positive advanced breast cancer
* Age>18 years.
* 1 to 10 brain metastases confirmed by enhanced brain MRI
* KPS≥70
* Life expectancy of more than 12 weeks
* Prior therapy of oral dexamethasone not exceeding 16mg/d
* Time interval from prior therapy was more than 2 weeks, and evaluation of adverse events is no more than grade 1.
* Maximum diameter of intracranial metastases is less than 3cm measured by enhanced brain MRI(2-3mm)
* Prior endocrine therapy were allowed
* Anti-Her2 targeted treatment were allowed
* Screening laboratory values must meet the following criteria( and should be obtained within 28 days prior to registration):

Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L, Platelets≥ 90 x 109/L, Hemoglobin ≥ 90 g/L Aspartate aminotransferase/alanine aminotransferase (AST/ALT) ≤2.5 x ULN without liver metastasis,≤ 5 x ULN with liver metastases Serum BUN and creatinine ≤ 1.5 x Upper Limit of Normal (ULN)

* Time interval from chemotherapy was more than 2 weeks, endocrine therapy and anti-Her2 targeted treatment are allowed to be used concurrently with FSRT
* Signed the informed consent form prior to patient entry

Exclusion Criteria:

* Leptomeningeal or hemorrhagic metastases
* Uncontrolled epilepsy
* Severe complication: cardiovascular disease, end-stage renal disease, severe hepatic disease, infection etc.
* Pregnancy or lactation period， women of child-bearing age who are unwilling to accept contraceptive measures.
* Inability to complete enhanced MRI
* Patients who are difficult or unable to be followed-up
* Not suitable for inclusion for specific reasons judged by sponsor
* Patients who are receiving cytotoxic drug concomitantly
* Have received prior radiotherapy for brain metastasis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
intracranial local tumor control rate | 2 years

SECONDARY OUTCOMES:
Intracranial distant metastasis rate | 2 years
  intracranial distant metastasis after FSRT will be determined by the development of intracranial distant metastasis is determined by new lesions outside of the irradiated area.
Intracranial Progression-Free Survival (PFS) | 2 years
  Time from the date of radiotherapy to the investigator-determined date of progression or death due to any cause, whichever occurs first
overall survival(OS) | 3 years
  time from the date of informed consent until to the date of death, regardless of the cause of death.
Adverse events | 2 years
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0.3

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No